CLINICAL TRIAL: NCT00882115
Title: Broccoli Sprout Extract Effects on the Inflammatory Response to Diesel Exhaust Particles in the Nose
Brief Title: Broccoli Sprout Extract Effects on Allergic Inflammation in the Nose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Professor of Clinical Medicine, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DAIT AADCRC-UCLA-01
Record Dates: First submitted 2009-04-14; First posted 2009-04-16 (Estimated); Results first posted 2018-11-15 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Allergic Airway Disease
Keywords: DEP; Broccoli Sprout Extract; Allergies
MeSH Terms: conditions — Hypersensitivity | interventions — sulforaphane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DEP challenge in subjects consuming BSE (Experimental): DEP will be administered in nostrils of participants who received BSE intervention by drinking 1 cup of liquid containing 1.25 g BSE daily for 4 days, or without consuming BSE.
  Interventions: Drug: Broccoli sprout extract (BSE)

INTERVENTIONS:
Drug: Broccoli sprout extract (BSE) — BSE will be ingested by drinking a liquid formula containing 1.25 g BSE in a volume equaling 1 cup daily for 4 consecutive days in the BSE intervention phase.
  Other Names: Sulforaphane

SUMMARY:
Allergic airway disease is a term used to describe conditions such as allergic rhinitis and asthma. Among other causative agents, air pollutants and diesel exhaust in particular, have been shown to create and also worsen existing allergic airway disease. These inhaled pollution particles have oxidative properties that drive inflammation-related effects through specific metabolic-associated processes. These processes are not adequately suppressed by current therapeutics. The purpose of this study is to explore the effects of broccoli sprout extract on the inflammatory process in the nose caused by diesel exhaust particles, which are important elements in air pollution. Broccoli sprout extract is a very potent inducer of Phase II enzymes (natural antioxidants).

DETAILED DESCRIPTION:
Antioxidant enzymes are proteins produced by the body to protect cells against the harmful effects of chemicals, such as those found in air pollution. Particulate air pollution and diesel exhaust in particular have been shown to cause and also exacerbate allergic airway disease. While there are ongoing efforts to improve air quality, there remains a need for alternative methods to address and prevent the adverse health effects of ambient air pollution, such as allergic rhinitis,, asthma, chronic obstructive pulmonary disease, and lung cancer. Currently, there are no therapeutic options which, directly target and address the effects of air pollutants in susceptible populations.

The purpose of this study is to examine the effect of broccoli sprout extract on airway inflammation caused by diesel exhaust particles. This study will analyze whether broccoli sprout extract will increase the levels of the natural, helpful, antioxidant enzymes in the nose and as a result decrease the inflammation caused by nasal exposure to diesel exhaust particles.

Participants will attend up to ten clinical visits, which include three screening visits. Some visits (2, 4, and 9) will last approximately 1 hour and require that the participants return to the clinic after 6 hours. The remaining visits (excluding Visit 1, which will also last about 1 hour) will take less than 30 minutes. Participants are restricted from consuming certain vegetables three days prior to, and during the course of the study.

During the screening phase, which will last from 4-5 days, and after giving informed consent participants will undergo a baseline evaluation that includes a medical history, a physical exam, blood drawing, allergy skin testing, nose washing, and a diesel exhaust particle (DEP) challenge test. For the DEP test, a small amount of fluid containing DEP particles will be sprayed in the nose (this amount is equivalent to the DEP that one breathes in over 2 days in Los Angeles). Investigators will also screen for natural antioxidant-related genes antioxidant enzymes and other indicators of DEP sensitivity. Female participants of child bearing potential will have a urine pregnancy test.

Participants will be asked to drink broccoli sprout extract for four days in a row (visits 6, 7, 8, and 9). The dosage is less than 1 cup and requires that participants fast 2 hours before the study visits when broccoli sprout extract is ingested. This study requires that participants be allergic to cat. An allergy skin test will be performed to determine whether they have this kind of allergy.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide informed consent
* DEP responder as defined in protocol
* Ability to refrain from consuming cruciferous vegetables 3 days prior to starting study and while on study. Cruciferous vegetables include: Broccoli, Kale, Chard, Kohlrabi, Brussels Sprouts, Parsley, Watercress, Daikon, Cabbage, Rutabagas, Cauliflower, Bok Choy, Arugula, Turnips, Radish, Mustard and Collard greens.
* Allergy skin test positive to cat
* Nonsmoker or ex-smoker of more than one year

Exclusion Criteria:

* Smoking within past year or during study
* Systemic corticosteroid or other immunosuppressive medication use in the previous 3 months or during study
* Intranasal corticosteroid use in the previous month or during the study
* Intranasal antihistamine or cromolyn use in the previous week or during study
* Allergen immunotherapy during the previous 12 months or during study
* Omalizumab use in the previous 12 months or during study
* Systemic antihistamine or leukotriene modifying medication use in the previous week or during study
* History of asthma or any current medical condition that in the opinion of the investigator may compromise the subject's ability to safely participate in the study
* Baseline abnormality of hemoglobin, platelets, leukocytes, serum chemistries, liver function testing, or presence of proteinuria
* A finding during physical examination that, in the opinion of the investigator may compromise the participant's ability to safely participate in the study
* Pregnant or breast-feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-07-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Heber, MD, PhD, Study Chair — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers.

REFERENCES:
- [Background] Krewski D. Evaluating the effects of ambient air pollution on life expectancy. N Engl J Med. 2009 Jan 22;360(4):413-5. doi: 10.1056/NEJMe0809178. No abstract available. PMID 19164194
- [Background] Munday R, Mhawech-Fauceglia P, Munday CM, Paonessa JD, Tang L, Munday JS, Lister C, Wilson P, Fahey JW, Davis W, Zhang Y. Inhibition of urinary bladder carcinogenesis by broccoli sprouts. Cancer Res. 2008 Mar 1;68(5):1593-600. doi: 10.1158/0008-5472.CAN-07-5009. Epub 2008 Feb 29. PMID 18310317
- [Background] Parker JD, Akinbami LJ, Woodruff TJ. Air pollution and childhood respiratory allergies in the United States. Environ Health Perspect. 2009 Jan;117(1):140-7. doi: 10.1289/ehp.11497. Epub 2008 Sep 30. PMID 19165401
- [Background] Pope CA 3rd, Ezzati M, Dockery DW. Fine-particulate air pollution and life expectancy in the United States. N Engl J Med. 2009 Jan 22;360(4):376-86. doi: 10.1056/NEJMsa0805646. PMID 19164188
- [Result] Heber D, Li Z, Garcia-Lloret M, Wong AM, Lee TY, Thames G, Krak M, Zhang Y, Nel A. Sulforaphane-rich broccoli sprout extract attenuates nasal allergic response to diesel exhaust particles. Food Funct. 2014 Jan;5(1):35-41. doi: 10.1039/c3fo60277j. PMID 24287881

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment period was 07/10/2009 - 11/09/2010. Enrollment took place in a private setting in the clinic located at the site.
Pre-assignment Details: Thirty-eight participants who tested positive for cat allergy were enrolled. The study had three phases: screen, control and intervention. There was a 2-week run in and a 4-week wash out period. Six subjects who did not respond to DEP challenge at screen phase, and three subjects who withdrew from the study before intervention were excluded.
Groups:
- Cell Count Change in Response to Nasal DEP Challenge.: Nasal cell count change in response to DEP challenge (300 microgram DEP in 200 microliter saline) in participants who received BSE by drinking 1 cup of liquid containing 1.25 g BSE daily for 4 days, or without consuming BSE.
Period: Overall Study
Arm/Group | Cell Count Change in Response to Nasal DEP Challenge.
Started | 38
Completed | 29
Not Completed | 9
Not completed — Withdrawal by Subject | 3
Not completed — did not respond to DEP challe | 6

BASELINE CHARACTERISTICS:
Groups:
- DEP Challenge in Subjects Consuming BSE: DEP will be administered in nostrils of participants who receive BSE by drinking 1 cup of liquid containing 1.25 g BSE daily for 4 days, or without consuming BSE.
Arm/Group | DEP Challenge in Subjects Consuming BSE
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Total Nasal Cell Count in Response to DEP Challenge at 0, 6 and 24 hr With or Without BSE Intervention
Description: Change of total nasal cell count in response to a standard diesel exhaust particle (DEP) challenge was determined by counting the total number of cells (leukocytes) recovered from nasal lavage fluid at 0 hr (just prior to DEP dosing), 6 hr and 24 hr later in participants who consuming BSE for 4 days, or without consuming BSE (control). Nasal challenges were performed with 300 microgram a standard DEP in 200 microliter saline.
Time Frame: 0, 6 and 24 hours at Control visit and BSE visit (Day 4 of intervention)
Population: All participants with baseline (0 hr), and 6 hr and 24 hr post-baseline nasal cell count measurement.
Measure: Mean (Standard Deviation); unit: log cells/mL
Groups:
- Nasal DEP Challenge: All participants consumed 1.25 g BSE suspended in juice once a day for 4 consecutive days prior to dosing of 300 microg DEP in 200 microL saline
Arm/Group | Nasal DEP Challenge
Number analyzed (Participants) | 29
log cells/mL
  0 hr prior DEP dosing (control) | 4.44 (0.51)
  6 hr after DEP dosing (control) | 4.50 (0.56)
  24 hr after DEP dosing (control) | 4.73 (0.52)
  0 hr prior to DEP doising with BSE intervention | 4.70 (0.54)
  6 hr after DEP dosing with BSE intervention | 4.44 (0.51)
  24 hr after DEP dosing with BSE intervention | 4.57 (0.46)
Statistical Analysis 1: Comparison: Nasal DEP Challenge; Comparison was made to the 24 h minus baseline change in both control phase and intervention phase; Test type: Other; p < 0.001, ANOVA; Data followed the normal distribution, therefore, a parametric repeated measure (mixed model) ANOVA model was used to compare means
Statistical Analysis 2: Comparison: Nasal DEP Challenge; Comparison waws made to the 6 hour minus baseline change in both control phase and intervention phase; Test type: Other; p < 0.01, ANOVA; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a 6 week period
Description: Participants were monitored and questioned regarding the occurrence and nature of any adverse experiences.
Arm/Group | Cell Count Change in Response to Nasal DEP Challenge
Serious Adverse Events (participants affected / at risk) | 5/38
Other Adverse Events (participants affected / at risk) | 4/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cell Count Change in Response to Nasal DEP Challenge (N=38)
mild discomfort (Gastrointestinal disorders) | 5 (8)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cell Count Change in Response to Nasal DEP Challenge (N=38)
nasal irritation, running nose (Skin and subcutaneous tissue disorders) | 4 (7)

LIMITATIONS AND CAVEATS:
The study tested the hypothesis that sulforaphane in the broccoli sprout extract (BSE) will interfere in the generation of nasal inflammation by diesel exhaust particles (DEP) but more studies with larger sample size and more data are needed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No